CLINICAL TRIAL: NCT06986369
Title: Effects of Rivaroxaban on Vascular Endothelial Function and Circulating Endothelial Progenitor Cells in Patients With Stable Atherosclerotic Vascular Diseases
Brief Title: Effects of Rivaroxaban on Vascular FMD in Patients With Stable Atherosclerotic Vascular Diseases
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Tse Hung Fat, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW 20-312
Record Dates: First submitted 2024-03-07; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Atherosclerosis, Coronary
MeSH Terms: conditions — Coronary Artery Disease | interventions — Rivaroxaban; Tablets

STUDY DESIGN:
Intervention Model Description: rivaroxaban and aspirin versus aspirin alone
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- rivaroxaban 2.5mg twice daily and aspirin 100mg once daily (Active Comparator): Rivaroxaban 2.5mg twice daily Oral Tablet novel oral anticoagulants , 2.5mg twice daily for 3 months and Aspirin 100 MG Oral Tablet, Enteric Coated antiplatelet agent, 100mg once daily for 3 months
  Interventions: Drug: Rivaroxaban 2.5 MG Oral Tablet [Xarelto]
- Aspirin 100mg daily for 3 months (No Intervention): Aspirin 100 MG Oral Tablet, Enteric Coated antiplatelet agent, 100mg once daily for 3 months

INTERVENTIONS:
Drug: Rivaroxaban 2.5 MG Oral Tablet [Xarelto] — prospective, randomized, 3 months study to clarify the efficacy of rivaroxaban and aspirin versus aspirin in the alone the changes on the number of circulating endothelial cells and endothelial function, and systemic inflammation, platelet and coagulation activation in patients with stable atherosclerotic vascular diseases.
  Other Names: Xarelto
  Arms: rivaroxaban 2.5mg twice daily and aspirin 100mg once daily

SUMMARY:
The specific mechanistic benefit of rivaroxaban versus other FXa inhibitors on atherothrombotic events remain unclear. Therefore plan to initiate a prospective, randomized study to investigate the effect of rivaroxaban and aspirin versus aspirin alone on changes of number circulating endothelial cells and endothelial function, and alteration in systemic inflammation, platelet and coagulation activation in patients with stable atherosclerotic vascular diseases.

The working hypothesis of this trial is that rivaroxaban and aspirin is superior to aspirin alone improvement in the number of circulating endothelial cells and endothelial function, assessed by flow-mediated vasodilatation, and reduction in systemic inflammation, platelet and coagulation activation in patients with stable atherosclerotic vascular diseases at 3 months follow-up.

DETAILED DESCRIPTION:
Factor Xa (FXa) and thrombin are well-known components of the coagulation cascade and other biological and pathophysiological processes that are linked to atherothrombotic as well as thromboembolic events. As a result, novel oral anticoagulants that are direct inhibitors of factor Xa (e.g., rivaroxaban) and thrombin (e.g.,dabigatran) have been developed for the prevention of thromboembolic recurrences in patients with venous thromboembolism and atrial fibrillation (AF) . Moreover, FXa inhibitors have also been investigated as an adjunct antithrombotic therapy in addition to dual antiplatelet therapy in selected patients with acute coronary syndrome. While APPRAISE-2 trial (apixaban), which was prematurely terminated because of an excess of bleeding and showed no evidence of benefit, ATLAS ACS 2 TIMI 51 trial (rivaroxaban) demonstrated a significant reduction in clinical events compared with placebo. These differences in clinical outcomes cannot be accounted by the discrepancy in the rates of bleeding, which was increased to a fairly similar extent in both trials. Moreover, recent clinical trials (COMPASS trial) in patients with stable atherosclerotic vascular diseases, either in patients with stable coronary artery disease (CAD) or peripheral artery disease (PAD), rivaroxaban plus aspirin reduced cardiovascular (CV) events but increased major bleeding compared with aspirin alone. Rivaroxaban alone did not differ from aspirin alone for CV events and increased major bleeding. Nevertheless, the specific mechanistic benefit of rivaroxaban versus other FXa inhibitors on atherothrombotic events remain unclear. During the development of atherosclerosis, vascular endothelial cells, platelets, pro-inflammatory cytokines and several serine proteases, such as thrombin, Xa and tissue factor can promote vascular inflammation and leukocyte infiltration via the activation of protease-activated receptor (PAR) signalling pathway. Indeed, FXa and thrombin mediated PAR activation contributes to the linking between coagulation and inflammatory pathways on the endothelium. In experimental studies, rivaroxaban showed a concentration-dependent positive effect on cell viability and growth of vascular endothelial cells verses controls. Furthermore, preclinical studies demonstrated that direct Xa inhibition can have anti-inflammatory and protective activities in atherosclerotic plaque development beyond anticoagulation.

Here, investigators hypothesize that the vascular protective effects of rivaroxaban are mediated via increasing endothelial progenitor cells and improvement of vascular endothelial function to reduce vascular inflammation and coagulation activation in patients with stable atherosclerotic vascular diseases.

ELIGIBILITY:
Inclusion Criteria:

patients must fulfill the following criteria.

* Willing and able to provide written informed consent
* CAD and/or PAD
* Subjects with CAD must also meet at least 1 of the following criteria:

Age 65 years or older, or Age younger than 65 years and documented atherosclerosis or revascularization involving at least 2 vascular beds or at least 2 additional risk factors:

* Current smoker (within 1 year of randomization)
* Diabetes mellitus
* Renal dysfunction with estimated glomerular filtration rate < 60 mL/min
* Heart failure
* Non-lacunar ischemic stroke >/= 1 month ago

Exclusion Criteria:

* High risk of bleeding
* Stroke within 1 month or any history of hemorrhagic or lacunar stroke
* Severe heart failure with known ejection fraction < 30% or New York Heart Association class III or IV symptoms
* Estimated glomerular filtration rate < 15 mL/min
* Need for dual antiplatelet therapy, other non-aspirin antiplatelet therapy, or oral anticoagulant therapy
* Known non-cardiovascular disease that is associated with poor prognosis (eg, metastatic cancer) or that increases the risk of an adverse reaction to study interventions
* History of hypersensitivity or known contraindication for rivaroxaban, aspirin, pantoprazole, or excipients, if applicable
* Systemic treatment with strong inhibitors of CYP3A4 as well as p-glycoprotein (eg, systemic azole antimycotics, such as ketoconazole, and HIV-protease inhibitors, such as ritonavir), or strong inducers of CYP 3A4 (ie, rifampicin, rifabutin, phenobarbital, phenytoin, and carbamazepine)
* Any known hepatic disease associated with coagulopathy
* Subjects who are pregnant, breastfeeding, or are of childbearing potential, and sexually active and not practicing an effective method of birth control (eg, surgically sterile, prescription oral contraceptives, contraceptive injections, intrauterine device, double- barrier method, contraceptive patch, male partner sterilization)
* Previous assignment to treatment during this study
* Concomitant participation in another study with investigational drug
* Known contraindication to any study-related procedures

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Endothelial Function | 3 months
  The Flow mediated dilatation of brachial artery at the baseline and the 3 months after randomization. Demonstrate brachial diameters, the measurement will be presented in absolute FMD millimeter (FMDmm). The report value should be present in FMD percentage (FMD%) as the mean of baseline measurement minus the mean of 3 months measurement then divided by the 3 months measurement.

SECONDARY OUTCOMES:
Plasma Adenosine Level Platelet Function Parameter Endothelial Progenitor Cell Count Biomarkers such as Highly Sensitive Troponin. | 3 months
  Collect the blood sample to test the Plasma adenosine level Platelet Function parameters Endothelial progenitor cell count biomarkers such as highly sensitive troponin at the baseline and 3 months after randomization. The unit of the test should be nmol/L.
Platelet function parameter and Coagulation parameter | 3 months
  VerifyNow test results were expressed in Aspirin Reaction Units (ARU) and LTA test results in percent of maximal aggregation. The cut-off for determination of aspirin resistance was > or =550 ARU and > or =20%, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Hung Fat Tse, Principal Investigator — Queen Mary Hospital, Hong Kong
Locations (1):
- Queen Mary Hospital, the University of Hong Kong, Hong Kong, China

REFERENCES:
- [Background] Borissoff JI, Spronk HM, ten Cate H. The hemostatic system as a modulator of atherosclerosis. N Engl J Med. 2011 May 5;364(18):1746-60. doi: 10.1056/NEJMra1011670. No abstract available. PMID 21542745
- [Background] Spronk HM, de Jong AM, Crijns HJ, Schotten U, Van Gelder IC, Ten Cate H. Pleiotropic effects of factor Xa and thrombin: what to expect from novel anticoagulants. Cardiovasc Res. 2014 Mar 1;101(3):344-51. doi: 10.1093/cvr/cvt343. Epub 2014 Jan 2. PMID 24385341
- [Background] Esmon CT. Targeting factor Xa and thrombin: impact on coagulation and beyond. Thromb Haemost. 2014 Apr 1;111(4):625-33. doi: 10.1160/TH13-09-0730. Epub 2013 Dec 12. PMID 24336942
- [Background] Eriksson BI, Quinlan DJ, Eikelboom JW. Novel oral factor Xa and thrombin inhibitors in the management of thromboembolism. Annu Rev Med. 2011;62:41-57. doi: 10.1146/annurev-med-062209-095159. PMID 21226611
- [Background] Alexander JH, Lopes RD, James S, Kilaru R, He Y, Mohan P, Bhatt DL, Goodman S, Verheugt FW, Flather M, Huber K, Liaw D, Husted SE, Lopez-Sendon J, De Caterina R, Jansky P, Darius H, Vinereanu D, Cornel JH, Cools F, Atar D, Leiva-Pons JL, Keltai M, Ogawa H, Pais P, Parkhomenko A, Ruzyllo W, Diaz R, White H, Ruda M, Geraldes M, Lawrence J, Harrington RA, Wallentin L; APPRAISE-2 Investigators. Apixaban with antiplatelet therapy after acute coronary syndrome. N Engl J Med. 2011 Aug 25;365(8):699-708. doi: 10.1056/NEJMoa1105819. Epub 2011 Jul 24. PMID 21780946
- [Background] Mega JL, Braunwald E, Wiviott SD, Bassand JP, Bhatt DL, Bode C, Burton P, Cohen M, Cook-Bruns N, Fox KA, Goto S, Murphy SA, Plotnikov AN, Schneider D, Sun X, Verheugt FW, Gibson CM; ATLAS ACS 2-TIMI 51 Investigators. Rivaroxaban in patients with a recent acute coronary syndrome. N Engl J Med. 2012 Jan 5;366(1):9-19. doi: 10.1056/NEJMoa1112277. Epub 2011 Nov 13. PMID 22077192
- [Background] Eikelboom JW, Connolly SJ, Bosch J, Dagenais GR, Hart RG, Shestakovska O, Diaz R, Alings M, Lonn EM, Anand SS, Widimsky P, Hori M, Avezum A, Piegas LS, Branch KRH, Probstfield J, Bhatt DL, Zhu J, Liang Y, Maggioni AP, Lopez-Jaramillo P, O'Donnell M, Kakkar AK, Fox KAA, Parkhomenko AN, Ertl G, Stork S, Keltai M, Ryden L, Pogosova N, Dans AL, Lanas F, Commerford PJ, Torp-Pedersen C, Guzik TJ, Verhamme PB, Vinereanu D, Kim JH, Tonkin AM, Lewis BS, Felix C, Yusoff K, Steg PG, Metsarinne KP, Cook Bruns N, Misselwitz F, Chen E, Leong D, Yusuf S; COMPASS Investigators. Rivaroxaban with or without Aspirin in Stable Cardiovascular Disease. N Engl J Med. 2017 Oct 5;377(14):1319-1330. doi: 10.1056/NEJMoa1709118. Epub 2017 Aug 27. PMID 28844192
- [Background] Connolly SJ, Eikelboom JW, Bosch J, Dagenais G, Dyal L, Lanas F, Metsarinne K, O'Donnell M, Dans AL, Ha JW, Parkhomenko AN, Avezum AA, Lonn E, Lisheng L, Torp-Pedersen C, Widimsky P, Maggioni AP, Felix C, Keltai K, Hori M, Yusoff K, Guzik TJ, Bhatt DL, Branch KRH, Cook Bruns N, Berkowitz SD, Anand SS, Varigos JD, Fox KAA, Yusuf S; COMPASS investigators. Rivaroxaban with or without aspirin in patients with stable coronary artery disease: an international, randomised, double-blind, placebo-controlled trial. Lancet. 2018 Jan 20;391(10117):205-218. doi: 10.1016/S0140-6736(17)32458-3. Epub 2017 Nov 10. PMID 29132879
- [Background] Anand SS, Bosch J, Eikelboom JW, Connolly SJ, Diaz R, Widimsky P, Aboyans V, Alings M, Kakkar AK, Keltai K, Maggioni AP, Lewis BS, Stork S, Zhu J, Lopez-Jaramillo P, O'Donnell M, Commerford PJ, Vinereanu D, Pogosova N, Ryden L, Fox KAA, Bhatt DL, Misselwitz F, Varigos JD, Vanassche T, Avezum AA, Chen E, Branch K, Leong DP, Bangdiwala SI, Hart RG, Yusuf S; COMPASS Investigators. Rivaroxaban with or without aspirin in patients with stable peripheral or carotid artery disease: an international, randomised, double-blind, placebo-controlled trial. Lancet. 2018 Jan 20;391(10117):219-229. doi: 10.1016/S0140-6736(17)32409-1. Epub 2017 Nov 10. PMID 29132880
- [Background] Alvarez E, Paradela-Dobarro B, Raposeiras-Roubin S, Gonzalez-Juanatey JR. Protective, repairing and fibrinolytic effects of rivaroxaban on vascular endothelium. Br J Clin Pharmacol. 2018 Feb;84(2):280-291. doi: 10.1111/bcp.13440. Epub 2017 Oct 25. PMID 28940408
- [Background] Lee IO, Kratz MT, Schirmer SH, Baumhakel M, Bohm M. The effects of direct thrombin inhibition with dabigatran on plaque formation and endothelial function in apolipoprotein E-deficient mice. J Pharmacol Exp Ther. 2012 Nov;343(2):253-7. doi: 10.1124/jpet.112.194837. Epub 2012 Jul 25. PMID 22837011
- [Background] Borissoff JI, Otten JJ, Heeneman S, Leenders P, van Oerle R, Soehnlein O, Loubele ST, Hamulyak K, Hackeng TM, Daemen MJ, Degen JL, Weiler H, Esmon CT, van Ryn J, Biessen EA, Spronk HM, ten Cate H. Genetic and pharmacological modifications of thrombin formation in apolipoprotein e-deficient mice determine atherosclerosis severity and atherothrombosis onset in a neutrophil-dependent manner. PLoS One. 2013;8(2):e55784. doi: 10.1371/journal.pone.0055784. Epub 2013 Feb 7. PMID 23409043
- [Background] Ragosta M, Gimple LW, Gertz SD, Dunwiddie CT, Vlasuk GP, Haber HL, Powers ER, Roberts WC, Sarembock IJ. Specific factor Xa inhibition reduces restenosis after balloon angioplasty of atherosclerotic femoral arteries in rabbits. Circulation. 1994 Mar;89(3):1262-71. doi: 10.1161/01.cir.89.3.1262. PMID 8124815
- [Background] Borissoff JI, Heeneman S, Kilinc E, Kassak P, Van Oerle R, Winckers K, Govers-Riemslag JW, Hamulyak K, Hackeng TM, Daemen MJ, ten Cate H, Spronk HM. Early atherosclerosis exhibits an enhanced procoagulant state. Circulation. 2010 Aug 24;122(8):821-30. doi: 10.1161/CIRCULATIONAHA.109.907121. Epub 2010 Aug 9. PMID 20697022